CLINICAL TRIAL: NCT03091257
Title: An Open-label, Pilot Study of Dabrafenib and/or Trametinib in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Dabrafenib and/or Trametinib in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry); Multiple Myeloma Research Consortium (Network); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Noopur Raje, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-352
Record Dates: First submitted 2017-02-17; First posted 2017-03-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dabrafenib (Experimental): Determine if mutation in BRAF, KRAS, NRAS
  * BRAF V600 mutated
  * Treat cohort with Dabrafenib
  * Analysis
  * Treat cohort with Dabrafenib
  Interventions: Drug: Dabrafenib
- Dabrafenib and Trametinib (Experimental): Determine if mutation in BRAF, KRAS, NRAS
  * BRAF V600 mutated, BRAF/KRAS mutated, or BRAF/NRAS mutated, or BRAF non-V600 mutated
  * Treat cohort with Dabrafenib and Trametinib
  * Analysis
  * Treat cohort with Dabrafenib and Trametinib
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Trametinib (Experimental): Determine if mutation in BRAF, KRAS, NRAS
  * KRAS or NRAS mutated
  * Treat cohort with Trametinib
  * Analysis
  * Treat cohort with Trametinib
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Administered Orally BID
  Other Names: Tafinlar
  Arms: Dabrafenib; Dabrafenib and Trametinib
Drug: Trametinib — Administered Orally once daily
  Other Names: Mekinist
  Arms: Dabrafenib and Trametinib; Trametinib

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for multiple myeloma.

The names of the study drugs involved in this study are:

* Trametinib
* Dabrafenib

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study drug in this disease. "Investigational" means that the combination of drugs is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved the drugs for your type of cancer.

The FDA has not approved Trametinib or Dabrafenib for your specific disease but they have been approved for other uses.

Some cancers have changes (mutations) in a gene called BRAF or other genes, called KRAS or NRAS. These three genes tell the body to make a protein called BRAF, KRAS, or NRAS, respectively, which are all involved in sending signals in cells that can lead to cell growth. Certain mutations in these three genes cause a change in these proteins that can increase the growth and spread of cancer cells.

Dabrafenib and trametinib work to prevent these altered proteins from working and sending signals in cancer cells, and thereby may block the growth and spread of cancer cells in people with cancers with BRAF, KRAS, or NRAS gene mutations. Dabrafenib and trametinib have been used in the treatment for other cancers in other research studies, and information from those research studies suggest that these agents may help to kill multiple myeloma cells.

Dabrafenib and trametinib, which are investigated in this research study may or may not kill myeloma cells effectively. We would like to see if these drugs given alone or in combination safely and effectively kill these cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of multiple myeloma as defined by the following criteria:

  * Monoclonal plasma cells in the bone marrow greater than or equal to 10% and/or presence of a biopsy-proven plasmacytoma
  * Monoclonal protein present in the serum and/or urine
  * Measurable disease as defined by the following:

    * IgG multiple myeloma: Serum monoclonal paraprotein (M-protein) level greater than or equal to 0.5 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours
    * IgA multiple myeloma: Serum M-protein level greater than or equal to 0.5 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours
    * IgD multiple myeloma: Serum M-protein level greater than or equal to 0.5 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours
    * Light chain multiple myeloma: Serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Participants must have myeloma that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains. Measurable disease is defined as one or more of the following: serum M-protein ≥0.5 g/dL, urine M-protein ≥200 mg/24 h, and/or serum FLC assay: involved FLC level ≥10 mg/dL with abnormal serum FLC ratio.
* Relapsed disease after at least 2 line of therapy
* Age ≥ 18 years years at the time of signing the informed consent form.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have sufficient organ and marrow function as defined below:

  * Participants with platelet level ≥50,000/mm3, within 21 days of initiation of protocol therapy for patients in whom <50% of bone marrow nucleated cells are plasma cells; or platelet count ≥30,000/mm3 for participants in whom >50% of bone marrow nucleated cells are plasma cells. Transfusion within 7 days of screening is not allowed to meet platelet eligibility criteria.
  * Participants with an absolute neutrophil count (ANC) ≥1000/mm3, within 21 days of initiation of protocol therapy. Growth factor within 7 days of screening is not allowed to meet ANC eligibility criteria.
  * Participants with hemoglobin level ≥ 8 g/dL, within 21 days of initiation of protocol therapy. Transfusion may be used to meet hemoglobin eligibility criteria.
  * Hepatic impairment, defined as total bilirubin ≤ 1.5 x institutional ULN (patients with benign hyperbilirubinemia (e.g., Gilbert's syndrome) are eligible.) or AST (SGOT), or ALT (SGPT), or alkaline phosphatase ≤ 2 x institutional ULN, within 21 days of initiation of protocol therapy.
  * PT/INR and PTT ≤ 1.3 x institutional upper limit of normal. Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to alternate assignment.
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal, except subjects with known Gilbert's syndrome.
  * Creatinine ≤ 2.0 mg/dl
  * Serum calcium or albumin-adjusted serum calcium ≥ 2.0 mmol/L (8.0 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL)
  * Left Ventricular Ejection Fraction (LVEF) ≥ LLN by ECHO. --- Abbreviations: ALT = alanine transaminase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; INR = international normalized ratio; LLN = lower limit of normal; PT = prothrombin time; PTT = partial thromboplastin time;
* Harboring a mutation in the BRAF oncogene or the KRAS or the NRAS oncogene
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to enrollment and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. A pregnancy test is not required for female participants over age 60 who have been postmenopausal for at least 24 months. Male participants, even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Ability to understand and the willingness to sign a written informed consent document.
* Participant must be able to swallow pills and retain oral medication and must not have clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.

Exclusion Criteria:

* Prior treatment with a BRAF inhibitor or a MEK inhibitor. Treatment by localized radiotherapy is not an exclusion criterion if an interval of at least two weeks between the end of radiotherapy and initiation of protocol therapy is observed.
* Primary amyloidosis (AL) or myeloma complicated by amyloidosis
* Nonsecretory multiple myeloma based upon standard M-component criteria (ie, measurable serum/urine M-component) unless the baseline serum free light chain level is elevated. Patients with plasmacytomas with biopsy proven known mutations may be included as long as they have evaluable disease by imaging.
* Participants receiving any other investigational agents within 2 weeks of the start of this trial and throughout the duration of this trial. Participants receiving anti-cancer treatment (chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment) within 3 weeks prior to first dose of dabrafenib or trametinib. Participants receiving proteasome inhibitors or immunomodulatory drugs (-imid), or chemotherapy without delayed toxicity within 2 weeks prior to first dose of dabrafenib or trametinib. Treatment by localized radiotherapy is not an exclusion criterion if an interval of at least two weeks between the end of radiotherapy and initiation of protocol therapy is observed.
* Current use of a prohibited medication as described in Section 6.4.
* Participants with platelet level <50,000/mm3, within 21 days of initiation of protocol therapy for patients in whom <50% of bone marrow nucleated cells are plasma cells; or platelet count <30,000/mm3 for participants in whom >50% of bone marrow nucleated cells are plasma cells. Transfusion within 7 days of screening is not allowed to meet platelet eligibility criteria.
* Participants with an absolute neutrophil count (ANC) <1000/mm3, within 21 days of initiation of protocol therapy. Growth factor within 7 days of screening is not allowed to meet ANC eligibility criteria.
* Participants with hemoglobin level < 8 g/dL, within 21 days of initiation of protocol therapy. Transfusion may be used to meet hemoglobin eligibility criteria.
* Hepatic impairment, defined as total bilirubin > 1.5 x institutional ULN (patients with benign hyperbilirubinemia (e.g., Gilbert's syndrome) are eligible.) or AST (SGOT), or ALT (SGPT), or alkaline phosphatase > 2 x institutional ULN, within 21 days of initiation of protocol therapy.
* Renal insufficiency, defined as serum creatinine >2.0 mg/dL.
* Participant had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class II, III or IV heart failure (see Appendix G), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities, or treatment refractory hypertension defined as a blood pressure of systolic >140mmHg and/ or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* A history or evidence of cardiovascular risk including any of the following:

  * A QT interval corrected for heart rate using the Bazett's formula (QTcB; Appendix E) ≥ 480 msec;
  * A history or evidence of current clinically significant uncontrolled arrhythmias; Clarification: Subjects with atrial fibrillation controlled for >30 days prior to dosing are eligible.
  * A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to alternate assignment.
  * A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines (Appendix G);
  * Patients with intra-cardiac defibrillators;
  * Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
  * Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy;
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
* A history of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and/or HCV will be permitted.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy or subjects with indolent second malignancies.
* Female participants pregnant or breast-feeding. Pregnant women are excluded from this study because dabrafenib, and trametinib may have teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued if the mother is treated with the study drugs. Dabrafenib was teratogenic and embryotoxic in rats at doses three times greater than the human exposure at the recommended clinical dose.
* A history or current evidence of retinal vein occlusion (RVO)
* History of interstitial lung disease or pneumonitis
* Patients with known human immunodeficiency virus (HIV) on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib and trametinib. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 100 weeks
  Response rate by IMWG criteria

SECONDARY OUTCOMES:
Number of Participants with Severe Adverse Events | 100 weeks
  NCI Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Noopur S Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No